CLINICAL TRIAL: NCT02326181
Title: Effects of Inspiratory and Respiratory Pressure Threshold Training in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effects of Inspiratory and Expiratory Pressure Training Methods in Patients With Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZJH21400964
Record Dates: First submitted 2014-12-21; First posted 2014-12-25 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Obstructive Pulmonary Disease(COPD)
Keywords: respiratory muscle training; respiratory muscle strength; respiratory endurance test; 6-minute walking test
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- control group (No Intervention): without inspiratory and expiratory pressure threshold training
- inspiratory pressure training group (Experimental): The patients will perform daily in 2 sessions of 30 minutes, using a pressure threshold trainer.
  Interventions: Device: inspiratory pressure training group
- mixed training group (Experimental): The patients will perform daily in 2 sessions of 30 minutes, using a pressure threshold trainer.
  Interventions: Device: mixed training group

INTERVENTIONS:
Device: inspiratory pressure training group — The respiratory pressure load device can be provided different loads to perform inspiratory and expiratory pressure training.In the study,pressure-threshold respiratory trainers were calibrated to provide different loads against inspiration (IMST) .
  Arms: inspiratory pressure training group
Device: mixed training group — The respiratory pressure load device can be provided different loads to perform inspiratory and expiratory pressure training.In the study,pressure-threshold respiratory trainers were calibrated to provide different loads against inspiration (IMST) and expiration(EMST).
  Arms: mixed training group

SUMMARY:
The study will investigate the effects of different training types ,including combined inspiratory with expiratory pressure threshold training,inspiratory pressure threshold training on patients with chronic obstructive airway disease and investigate whether expiratory pressure threshold training associated with inspiratory pressure threshold training would be better than inspiratory pressure threshold training alone, with regard to exercise capacity, respiratory muscle strength and endurance.

DETAILED DESCRIPTION:
We will study 60 patients diagnosed of chronic obstructive pulmonary disease.The monitoring will be done for 8 weeks. Pressure-threshold respiratory trainers were calibrated to provide different loads according to the patients against inspiration (IMST) or expiration (EMST). Those chronic obstructive pulmonary disease clinically stable patients stratified from mild to very severe GOLD stages, were blinded to randomly divided into 3 different groups: a)control group:without any training;b) inspiratory and expiratory pressure threshold training group: trained with the pressure threshold trainer twice time daily with 15minutes' duration;c)inspiratory pressure threshold training group:trained with the pressure threshold trainer twice time daily with 15 minutes' duration,different from the b group,the expiratory pressure threshold is calibrated at 0.

ELIGIBILITY:
Inclusion Criteria:

Clinically stable COPD with diagnosis of forced expiratory volume at one second(FEV1)/forced vital capacity(FVC) < 70%

Exclusion Criteria:

Cancer Unstable heart disease Neuromusculoskeletal disorder mental disorder Active smokers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
respiratory muscle strength measurements | baseline and 8 weeks

SECONDARY OUTCOMES:
respiratory muscle endurance text | baseline and 8 weeks
6-minute walking test | baseline and 12 weeks
perceived exertion for leg fatigue (Borg-scale) | baseline and 8 weeks
modified british medical research council(mMRC) questionnaire | baseline and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xin Chen, Doctor, Principal Investigator — Zhujiang Hospital
Locations (1):
- Zhujiang hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Xu W, Li R, Guan L, Wang K, Hu Y, Xu L, Zhou L, Chen R, Chen X. Combination of inspiratory and expiratory muscle training in same respiratory cycle versus different cycles in COPD patients: a randomized trial. Respir Res. 2018 Nov 20;19(1):225. doi: 10.1186/s12931-018-0917-6. PMID 30458805